CLINICAL TRIAL: NCT03580109
Title: Spa Therapy for Upper or Lower Limb Lymphoedema : a Randomized and Comparative Study
Brief Title: Spa Therapy for Upper or Lower Limb Lymphoedema
Acronym: THERMOEDEME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Association Francaise pour la Recherche Thermale (Other)
Collaborators: Floralis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: THERMOEDEME
Record Dates: First submitted 2018-06-05; First posted 2018-07-09 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Lymphoedema; Breast Cancer; Malignant Disease; Gynaecological Cancer; Lymphoma; Prostate Cancer
Keywords: Lymphoedema; Post breast cancer; Spa therapy; Education therapeutic; Malignant Disease; Post gynaecological cancer; Post Lymphoma; Post prostate cancer
MeSH Terms: conditions — Lymphedema; Breast Neoplasms; Lymphoma; Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: 2 groups:
  * Immediate spa therapy: the patient carries out the spa therapy with education therapeutic soon after the enrolment in the study
  * Late spa therapy: the patient carries out the spa therapy with education therapeutic after the 6-month follow up
Who Masked: Investigator
Masking Description: The investigator doesn't know the group of randomization of the patient. The spa therapy organisation is managed by the coordination center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate spa treatment (Active Comparator): Spa treatment linked with education therapeutic during 18 days just after randomization : common to all of spa resorts
  Interventions: Other: Immediate spa treatment
- Late spa treatment (Sham Comparator): Spa treatment linked with education therapeutic during 18 days 6 months visit after randomization
  Interventions: Other: Late spa treatment

INTERVENTIONS:
Other: Immediate spa treatment — Spa treatment linked education therapeutic in lymphoedema post breast cancer (whirlpool bath with automatic air and water massage cycles, massaging shower/individuals and groups educational sessions)
  Arms: Immediate spa treatment
Other: Late spa treatment — Spa treatment linked education therapeutic in lymphoedema post breast cancer (whirlpool bath with automatic air and water massage cycles, massaging shower/individuals and groups educational sessions)
  Arms: Late spa treatment

SUMMARY:
THERMOEDEME is a comparative, controlled, randomized, multicenter and simple blinded (investigator) trial.

The aim of this study is to evaluate effects of spa therapy in phlebology with a therapeutic education program in daily life of patients suffering lymphoedema.

DETAILED DESCRIPTION:
Lymphoedema is a chronic disease related to an insufficiency of the lymphatic system, which most often affects the limbs. Secondary forms are the most common, particularly those following surgical and radiotherapy treatments for cancer, the most classic being the post-therapeutic large arm of breast cancer.

The lymphoedema is a traditional phlebology indication in spa therapy. The spa therapy linked with therapeutic education could constitute a favorable environment for the treatment of lymphoedema.

The primary endpoint is the comparison of the rate of patients improved from baseline to 6 months on LMS27 (upper limb lymphoedema) or LYMQOL-LEG (lower limb lymphoedema) (Improvement is defined as 7 points between baseline and 6-month follow-up).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* available for a spa treatment (phlebology indication) during 18 days and a follow up period of 15 months
* with permanent lymphoedema of the upper or lower limb (2 ou 3 stade of International Society for Lymphology scale)
* voluntary to participate to the study, informed consent form signed after appropriate information
* affiliation to the social security system or equivalent

Exclusion Criteria:

* cancer undergoing chemotherapy and radiotherapy treatment in primary phase
* the baseline score of LMS27 or LYMQOL-LEG > 79
* pain of upper limb linked with a radical plexitis
* contra-indication of spa treatment (cancer in progress, psychiatrics disorders, immunodeficiency)
* Erysipelas case history in the last 6 months or pachyderma and lymphangiectasia
* no previous spa treatment for upper limb lymphoedema during the spa year
* risk of intensive treatment in the next 6 months
* subject participating to an other clinical study interventional
* pregnancy, parturient or breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evolution of lymphoedema quality of life assessed by the rate of patient with an improvement of the LMS27 scale (for upper limb lymphoedema). | 6 months
  Rate of patients with an improvement of 7 points minimum of the LMS27 scale (specific quality of life scale in upper limb lymphoedema) at 6 months.
  The LMS27 scale is composed of 27 questions with 5 answers possible : never, rarely, sometimes, often, always. The answer's score is respectively 1 (worse outcome) to 5 (better outcome). The higher the score is, the better the lymphoedema quality of life is.
Evolution of lymphoedema quality of life assessed by the rate of patient with an improvement of the LYMQOL-LEG scale (for lower limb lymphoedema). | 6 months
  Rate of patients with an improvement of 7 points minimum of the LYMQOL-LEG scale (specific quality of life scale in lower limb lymphoedema) at 6 months.
  The LYMQOL-LEG scale is composed of 26 questions with 4 answers possible: not at all, a little, quite a bit, a lot.
  In order to to standardize with the LMS27 scale (for upper limb lymphoedema), the quotations are reversed: the answer's score is respectively 1 (worse outcome) to 4 (better outcome). The higher the score is, the better the lymphoedema quality of life is.

SECONDARY OUTCOMES:
Evolution of lymphoedema quality of life assessed by the LMS27 scale (for upper limb lymphoedema) before / after spa therapy. | 6 and 12 months
  Evolution of the LMS27 scale (specific quality of life scale in upper limb lymphoedema) at 6 and 12 months.
  The LMS27 scale is composed of 27 questions with 5 answers possible : never, rarely, sometimes, often, always. The answer's score is respectively 1 (worse outcome) to 5 (better outcome). The higher the score is, the better the lymphoedema quality of life is.
Evolution of lymphoedema quality of life assessed by the LYMQOL-LEG scale (for lower limb lymphoedema) before / after spa therapy. | 6 and 12 months
  Evolution of the LYMQOL-LEG scale (specific quality of life scale in lower limb lymphoedema) at 6 and 12 months.
  The LYMQOL-LEG scale is composed of 26 questions with 4 answers possible: not at all, a little, quite a bit, a lot.
  In order to to standardize with the LMS27 scale (for upper limb lymphoedema), the quotations are reversed: the answer's score is respectively 1 (worse outcome) to 4 (better outcome). The higher the score is, the better the lymphoedema quality of life is.
Evolution of lymphoedema quality of life assessed by the most embarrassing items of the LMS27 scale (for upper lymphoedema). | 6 and 12 months
  Evolution of 5 items the most embarrassing chosen by the patients in the LMS27 scale (specific quality of life scale in upper limb lymphoedema) at 6 and 12 months.
  The LMS27 scale is composed of 27 questions with 5 answers possible : never, rarely, sometimes, often, always. The answer's score is respectively 1 (worse outcome) to 5 (better outcome). The higher the score is, the better the lymphoedema quality of life is.
Evolution of lymphoedema quality of life assessed by the most embarrassing items of the LYMQOL-LEG scale (for lower limb lymphoedema) | 6 and 12 months
  Evolution of 5 items the most embarrassing chosen by the patients in the LYMQOL-LEG scale (specific quality of life scale in lower limb lymphoedema) at 6 and 12 months.
  The LYMQOL-LEG scale is composed of 26 questions with 4 answers possible: not at all, a little, quite a bit, a lot.
  In order to to standardize with the LMS27 scale (for upper limb lymphoedema), we decide to reverse the quotations: the answer's score is respectively 1 (worse outcome) to 4 (better outcome). The higher the score is, the better the lymphoedema quality of life is.
Improvement of quality of life assessed by the generic quality of life: Euroquol EQ5D-3L | 6 and 12 months
  Improvement of generic quality of life (the Euroquol EQ5D-3L scale) at 6 and 12 months.
  EQ5D-3L is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of lige that can be used in a wide range of health conditions and treatments. The EQ5D-3L has 6 items intended to measure general health. The top 5 rate mobility, independence, daily activities, pain / discomfort, and anxiety / depression, and are rated according to 3 values from "No problem" to "Problem" or "Incapacity". This results in an index score. The last item deals with perceived health on the day the questionnaire is filled in and uses a visual analogue scale from 0 (wors) to 100 (best health possible) (Visual Analog Scale Score)
Upper or lower limb evaluation | 6 and 12 months
  Evolution of the volume of the upper or lower extremity evaluated (overall and then by segment) from staged perimeter measurements at 6 and 12 months.
Consumption of care between the 2 groups (immediate treatment/delayed treatment) | 6 and 12 months
  Evaluation of the costs incurred by lymphoedema (hospitalisations, medical and paramedical acts, treatments).
Compliance of spa therapy | After spa therapy
  Evaluation of the spa therapy compliance : number of health care performed in spa therapy.
Achievement educational aims | 3 months, 9 months.
  Verification of the achievement of educational targets in spa therapy by phone follow up.
Adverse events | 12 months
  Evaluation of all adverse events related to treatment, or not, according to the usual criteria of pharmacovigilance in clinical trials.
Functional evaluation | 12 months
  Monthly measurements of functional discomfort from inclusion to 12 months; The functional discomfort is measured monthly by a visual scale : not discomfort to maximal discomfort.
Long term evaluation | 12 months
  Evaluation of the maintenance of benefits at 12 months (stability of the long term effect) on the primary outcome and secondary outcomes.
Effect size | 6 and 12 months
  Confirmation of the extent of the effect between 6 and 12 months on the primary outcome and secondary outcomes.
Sub group analysis | 6 months
  Sub group analysis on the primary outcome measure (stratification on primo spa therapy, lymphoedema severity and lymphoedema localization)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick CARPENTIER, MD, Principal Investigator — Hospital University Grenoble
Locations (13):
- France (13):
  - Cabinet de médecine vasculaire, Albertville
  - CHU Amiens Picardie, Amiens
  - Thermes Argelès-Gazost, Argelès-Gazost
  - Thermes Barbotan Les Bains, Barbotan-les-Thermes
  - Groupe Hospitalier Mutualiste, Grenoble
  - Thermes La Léchère, La Léchère
  - CH Lourdes, Lourdes
  - Thermes Luz Saint Sauveur, Luz-Saint-Sauveur
  - Centre Léon Berard, Lyon
  - CH Tarbes, Tarbes
  - CHU Toulouse, Toulouse
  - Clinique générale HPDA, Valence
  - Clinique du Tonkin, Villeurbanne

REFERENCES:
- [Background] Rockson SG, Rivera KK. Estimating the population burden of lymphedema. Ann N Y Acad Sci. 2008;1131:147-54. doi: 10.1196/annals.1413.014. PMID 18519968
- [Background] International Society of Lymphology. The diagnosis and treatment of peripheral lymphedema. Consensus document of the International Society of Lymphology. Lymphology. 2003 Jun;36(2):84-91. PMID 12926833
- [Background] Carpentier PH, Blaise S, Satger B, Genty C, Rolland C, Roques C, Bosson JL. A multicenter randomized controlled trial evaluating balneotherapy in patients with advanced chronic venous insufficiency. J Vasc Surg. 2014 Feb;59(2):447-454.e1. doi: 10.1016/j.jvs.2013.08.002. Epub 2013 Oct 15. PMID 24135621
- [Background] Pusic AL, Cemal Y, Albornoz C, Klassen A, Cano S, Sulimanoff I, Hernandez M, Massey M, Cordeiro P, Morrow M, Mehrara B. Quality of life among breast cancer patients with lymphedema: a systematic review of patient-reported outcome instruments and outcomes. J Cancer Surviv. 2013 Mar;7(1):83-92. doi: 10.1007/s11764-012-0247-5. Epub 2012 Dec 5. PMID 23212603
- [Background] Norman GR, Sloan JA, Wyrwich KW. The truly remarkable universality of half a standard deviation: confirmation through another look. Expert Rev Pharmacoecon Outcomes Res. 2004 Oct;4(5):581-5. doi: 10.1586/14737167.4.5.581. PMID 19807551
- [Background] Norman GR, Sloan JA, Wyrwich KW. Interpretation of changes in health-related quality of life: the remarkable universality of half a standard deviation. Med Care. 2003 May;41(5):582-92. doi: 10.1097/01.MLR.0000062554.74615.4C. PMID 12719681
- [Background] Devoogdt N, Lemkens H, Geraerts I, Van Nuland I, Flour M, Coremans T, Christiaens MR, Van Kampen M. A new device to measure upper limb circumferences: validity and reliability. Int Angiol. 2010 Oct;29(5):401-7. PMID 20924341
- [Background] Lymphœdema Framework. Best Practice for the Management of Lymphœdema. International consensus. London: MEP Ltd, 2006:1-54.
- [Background] Vignes S. [Management of limb lymphedema]. Rev Med Interne. 2012 May;33(5):268-72. doi: 10.1016/j.revmed.2011.12.012. Epub 2012 Jan 31. French. PMID 22296831
- [Background] Carpentier PH, Fabry R. Crénothérapie des maladies vasculaires. In: Queneau P, editor. Médecine Thermale, faits et preuves. Paris: Masson Ed; 2000. p. 102-15.
- [Background] Carpentier PH, Colomb M, Poensin D, Satger B. [Incidence of erysipelas of the lower limbs in a spa resort. Efficacy of a strategy of sanitation education (La Lechere: 1992-1997)]. J Mal Vasc. 2001 Apr;26(2):97-9. French. PMID 11319415
- [Background] Blaise S, Villemur B, Richaud C, Rastel D, Bucci B, Evra V, Bouchet JY, les membres du réseau GRANTED, B.Satger. Conception d'un programme d'éducation thérapeutique pour les patients porteurs de lymphoedème : " Vivre avec un lymphoedème ". J Mal Vasc 2011,online access : doi:10.1016/j.jmv.2011.10.006
- [Background] Carpentier PH, Satger B, Poensin D, Trens C, Arnold M, Trolliet C, Noilhetas J, Chauvin E, Laurès J Therapeutic education combined with balneotherapy in lymphedema patients. Communication acceptée à l'American Venous Forum (Orlando 25/02/2016, publication en préparation)
- [Background] Launois R, Alliot F. Quality of Life Scale in Upper Limb Lymphoedema - A validation Study. Lymphology 33, 2000 (Suppl) : 266-74.
- [Background] Lim P, Li H, Neoh D, Ng SK. Health-related Quality of Life Measurement Tools for Lymphedema: A Review of the Literature. Plast Reconstr Surg Glob Open. 2022 Apr 27;10(4):e4276. doi: 10.1097/GOX.0000000000004276. eCollection 2022 Apr. PMID 37073384
- [Background] Keeley, Vaughan; Crooks, Sue; Locke, Jane; Veigas, Debbie; Riches, Katie and Hilliam, Rachel (2010). A quality of life measure for limb lymphoedema (LYMQOL). Journal of Lymphoedema, 5(1) pp. 26-37